CLINICAL TRIAL: NCT07223216
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BMF-650 in Otherwise Healthy Overweight or Obese Participants.
Brief Title: Study of BMF-650 in Otherwise Healthy Overweight or Obese Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biomea Fusion Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLP-131
Record Dates: First submitted 2025-10-29; First posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Obesity
Keywords: Obesity; Obsess; Overweight; Weight-loss; GLP-1; GLP-1 agonist; GLP-1 receptor agonist
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Intervention Model Description: This is a single center, double-blind, randomized, placebo-controlled, first-in-human (FIH) study of BMF-650, an oral non-peptide GLP-1 receptor agonist administered to otherwise healthy overweight or obese participants. Part 1 is a single ascending dose (SAD) study and Part 2 is a multiple ascending dose (MAD) study.
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study. Treatment assignment will not be known to the participants, the sponsor or the staff who are involved in the clinical evaluation of the participants and the analysis of data as indicated in the blinding plan. If appearance matching of the placebo is not possible then use of masking and/or unblinded dosing teams will be used to preserve the study blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part 1 SAD Cohort 1 (Regimen A) (Experimental): BMF-650 Tablets 10 mg or matching placebo in fasted state
  Interventions: Drug: BMF-650
- Part 1 SAD Cohort 2 (Regimen B and C) (Experimental): Regimen B:
  BMF-650 Tablets 25 mg or matching placebo in fasted state
  Regimen C:
  BMF-650 Tablets 25 mg or matching placebo in fed state (high-fat breakfast 30 minutes before BMF-650 or placebo is administered)
  Interventions: Drug: BMF-650
- Part 1 SAD Cohort 3 (Regimen D) (Experimental): BMF-650 Tablets 50 mg or matching placebo in fasted state
  Interventions: Drug: BMF-650
- Part 1 SAD Cohort 4 (Regimen E and F) (Optional) (Experimental): Regimen E:
  BMF-650 Tablets 100 mg or matching placebo in fasted state
  Regimen F:
  BMF-650 Tablets 100 mg or matching placebo in fed state (high-fat breakfast 30 minutes before BMF-650 or placebo is administered)
  Interventions: Drug: BMF-650
- Part 1 SAD Cohort 5 (Regimen G) (Optional) (Experimental): BMF-650 Tablets 200 mg or matching placebo in fasted state
  Interventions: Drug: BMF-650
- Part 2 MAD Cohort 1 (Regimen H) (Experimental): BMF-650 Tablets or matching placebo in fasted state
  10 mg QD for 7 days; 25 mg QD for 7 days; 50 mg QD for 7 days; 100 mg QD for 21 days.
  Interventions: Drug: BMF-650
- Part 2 MAD Cohort 2 (Regimen I) (Experimental): BMF-650 Tablets or matching placebo in fasted state
  25 mg QD for 7 days; 50 mg QD for 7 days; 100 mg QD for 7 days; 200 mg QD for 21 days.
  Interventions: Drug: BMF-650
- Part 2 MAD Cohort 3 (Regimen J) (Experimental): BMF-650 Tablets or matching placebo in fasted state
  25 mg QD for 7 days; 75 mg QD for 7 days; 150 mg QD for 7 days; 300 mg QD for 21 days.
  Interventions: Drug: BMF-650
- Part 2 MAD Cohort 4 (Regimen K) (Optional) (Experimental): BMF-650 Tablets or matching placebo in fasted state
  50 mg QD for 7 days; 100 mg QD for 7 days; 200 mg QD for 7 days; 400 mg QD for 21 days.
  Interventions: Drug: BMF-650

INTERVENTIONS:
Drug: BMF-650 — Interventional Product

SUMMARY:
A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BMF-650 in Otherwise Healthy Overweight or Obese Participants.

DETAILED DESCRIPTION:
This is a single center, double-blind, randomized, placebo-controlled, first-in-human (FIH) study of BMF-650, an oral non-peptide GLP-1 receptor agonist administered to otherwise healthy overweight or obese participants. Part 1 is a single ascending dose (SAD) study and Part 2 is a multiple ascending dose (MAD) study.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to understand a written informed consent, which must be obtained prior to initiation of study procedures.
2. Must be willing and able to comply with all study requirements
3. Healthy males or non-pregnant, non-lactating healthy females with obesity or overweight.
4. For Part 1 (SAD cohorts), BMI of 25.0 to 40.0 kg/m2 as measured at screening, with no chronic health conditions.
5. For Part 2 (MAD cohorts), BMI of 30.0 to 45.0 kg/m2, as measured at screening with no chronic health conditions.
6. Have a stable body weight (less than or equal to 5% body weight gain or loss) for 3 months prior to screening.
7. HbA1c ≤ 6.5%

Exclusion Criteria:

Medical/Surgical History and Mental Health

1. Known self or family history (first-degree relative) of medullary thyroid cancer and/or multiple endocrine neoplasia Type 2 (MEN2).
2. History of stomach or intestinal surgery or resection and/or gastroparesis (except that appendectomy and/or hernia repair will be allowed).
3. Significant history of or currently have major depressive disorder or psychiatric disorder or suicidal ideation within the last 2 years.
4. Severe uncontrolled treated or untreated hypertension (systolic blood pressure [BP] >150 mmHg or diastolic BP >90 mmHg).
5. Mean QTcF interval greater than 450 msec on triplicate ECGs.

   Diagnostic Assessments
6. Clinically significant abnormal clinical chemistry, hematology, coagulation or urinalysis as judged by the investigator
7. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) antibody results.
8. eGFR of <60 mL/min/1.73 m2
9. AST, ALT or total bilirubin > ULN
10. Lipase and/or amylase > ULN
11. Calcitonin ≥20 ng/L

    Prior Study Participation
12. Participants who have received any IMP in a clinical research study within 5 half -lives or within 30 days prior to first dose

    Prior and Concomitant Medication
13. Participants who are taking, or have taken, any prescribed or over-the-counter drug or herbal remedies (other than HRT/hormonal contraception) in the 14 days before first IMP administration
14. Use of prescription or over-the-counter medications known to significantly prolong the QT or QTc interval is excluded.
15. Currently dieting (formal weight loss program) and/or are currently using or have used within 2 months of screening any drugs for weight management
16. Participants who have previously used GLP-1 receptor agonist, or GIP/GLP-1 dual receptor agonists, or any investigational medicine containing a GLP-1 and/or GIP receptor agonist in the 6 months prior to first IMP administration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Assess safety and tolerability of BMF-650 | Time Frame:6 weeks (Part 1) and 11 weeks (Part 2)
  Incidence of adverse events (AEs)
Assess safety and tolerability of BMF-650 | Time Frame:6 weeks (Part 1) and 11 weeks (Part 2)
  Vital signs like blood pressure
Assess safety and tolerability of BMF-650 | Time Frame:6 weeks (Part 1) and 11 weeks (Part 2)
  ECG measures like QTcF interval
Assess safety and tolerability of BMF-650 | Time Frame:6 weeks (Part 1) and 11 weeks (Part 2)
  Physical examinations like general appearance
Assess safety and tolerability of BMF-650 | Time Frame:6 weeks (Part 1) and 11 weeks (Part 2)
  Safety labs like clinical chemistry

SECONDARY OUTCOMES:
Evaluate PK and food effect of BMF-650 in fed and fasted states | Time Frame:6 weeks (Part 1) and 11 weeks (Part 2)
  Tmax
Evaluate PK and food effect of BMF-650 in fed and fasted states | Time Frame:6 weeks (Part 1) and 11 weeks (Part 2)
  Cmax
Evaluate PK and food effect of BMF-650 in fed and fasted states | Time Frame:6 weeks (Part 1) and 11 weeks (Part 2)
  AUC(0-last)
Evaluate PK and food effect of BMF-650 in fed and fasted states | Time Frame:6 weeks (Part 1) and 11 weeks (Part 2)
  AUC(0-inf)
Evaluate PK and food effect of BMF-650 in fed and fasted states | Time Frame:6 weeks (Part 1) and 11 weeks (Part 2)
  T1/2

CONTACTS AND LOCATIONS:
Overall Officials: Biomea Fusion Inc., Study Director — Biomea Fusion Inc.
Locations (1):
- Medpace Clinical Pharmacology, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No